CLINICAL TRIAL: NCT04538352
Title: Transition From Basal/Bolus to Once-weekly Subcutaneous Semaglutide and Basal Insulin in Patients With Type-2 Diabetes Mellitus (TRANSITION-T2D) A Prospective Randomized Controlled Trial
Brief Title: Transition From Basal/Bolus to Once-weekly Subcutaneous Semaglutide and Basal Insulin in Patients With T2D
Acronym: TRANSITION-T2D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Kevin M Pantalone, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-853
Record Dates: First submitted 2020-08-29; First posted 2020-09-04 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; insulin degludec; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Once-weekly sc semaglutide combined with once-daily insulin (Experimental): Patients randomized to continue with MDI will be transitioned from their existing regimen to the rapid-acting insulin product insulin aspart and their basal insulin switched to once-daily insulin degludec.
  Interventions: Drug: Semaglutide; Drug: Insulin Degludec; Drug: Insulin aspart
- MDI requiring multiple daily injections of insulin (Experimental): Patients randomized to MDI will be allowed to continue correction rapid-acting insulin, in addition to their prandial doses of rapid-acting insulin, throughout the duration of the study.
  Interventions: Drug: Insulin Degludec; Drug: Insulin aspart

INTERVENTIONS:
Drug: Semaglutide — Medication for type 2 diabetes management
  Other Names: Ozempic
  Arms: Once-weekly sc semaglutide combined with once-daily insulin
Drug: Insulin Degludec — Medication for type 2 diabetes management
  Other Names: Tresiba
Drug: Insulin aspart — Medication for type 2 diabetes management (rapid-acting)
  Other Names: Novolog

SUMMARY:
This study is designed to determine whether therapy with once-weekly sc semaglutide in combination with once-daily insulin degludec will be capable of maintaining (or improving) glycemic control, when substituted for multiple daily injections of insulin (MDI), in patients with T2D with adequate glycemic control (≤ 7.5%) on MDI-based regimens (≤ 80 units of insulin per day), vs. further titration of insulin therapy in those continuing MDI. Weight loss, hypoglycemic episodes, and improvement in diabetes-treatment satisfaction will also be assessed between the two groups.

DETAILED DESCRIPTION:
Patients with type-2 diabetes mellitus (T2D) are often overweight or obese. In order to obtain adequate glycemic control, many of these patients require intensive therapy with multiple daily injections of insulin (referred to as MDI, basal/bolus regimen), using a rapid-acting/bolus insulin at each meal in combination with a once- or twice-daily long- acting/basal insulin. Unfortunately, intensive insulin therapy can result in undesired weight gain, which may, in part, result in further insulin resistance. In addition, weight gain may adversely affect the control of comorbid health conditions (hypertension, hyperlipidemia, congestive heart failure, sleep apnea, etc.). The burden of disease management with multiple daily injections of insulin also serves as a barrier to A1C goal attainment as maintaining compliance with such complex regimens is often challenging in the real-world setting.

Once patients with T2D require multiple daily injections of insulin to obtain glycemic control, it is generally considered to be a permanent/life-long therapy. However, reports have demonstrated the safety and effectiveness of adding once-daily glucagon-like peptide-1 receptor agonist (GLP-1RA) liraglutide to basal insulin therapy in order to obtain glycemic control (1, 2), and in clinical practice, the addition of liraglutide (or other FDA-approved GLP-1RAs) to basal insulin often negates or delays the need to initiate prandial insulin. Subsequently, a newer form of anti-diabetic therapy, a once-daily injectable combination of GLP-1RA and basal insulin, became available and demonstrated promise that perhaps glycemic control may even be obtained with less complex regimens (i.e., less daily injections). There are currently two GLP-1RA/basal insulin combination therapies that are FDA approved: iGlarLixi (Soliqua®), and iDegLira (Xultophy®) (3, 4). While these observations with iGlarLixi and iDegLira demonstrating an improvement in A1C while avoiding prandial insulin injections are very exciting, what remains unclear is if patients with reasonable glycemic control (A1C ≤ 7.5%) currently receiving MDI (basal/bolus, 3-4 injections per day) could potentially maintain or even improve glycemic control by switching to a once-daily injectable product like Xultophy® or Soliqua®. Currently, there are no studies available (or planned) that have answered this clinical question. One limitation of these combination products in the clinical setting is the inability to independently titrate the GLP-1RA and basal insulin components. If a patient begins to experience hypoglycemia, and/or their fasting BG values are currently within the goal range, the dose of these combination products cannot be further titrated, limiting one's ability to further improve glycemic control in patients with a residual A1C elevation.

What also remains unclear is if some of the newer formulations of GLP-1RA may also be able to reduce the burden of disease management and maintain glycemic control in patients who are currently well-controlled on a regimen of MDI. Recently, subcutaneous (sc) once-weekly semaglutide has been demonstrated to be capable of improving glycemic control in patients with T2D in combination with insulin therapy. In SUSTAIN-5 (5), at week 30, subcutaneous semaglutide 0.5 and 1.0 mg was demonstrated to reduce A1C by 1.4% and 1.8%, respectively, vs 0.1% with placebo [mean baseline A1C value, 8.4%] in a population of T2D patients receiving stable therapy with basal insulin with or without metformin. Moreover, mean body weight (kg) decreased with semaglutide 0.5 and 1.0 mg vs placebo from baseline to end of treatment: 3.7, 6.4, and 1.4 kg, respectively. Premature treatment discontinuation due to adverse events was higher for semaglutide 0.5 and 1.0 mg vs placebo (4.5%, 6.1%, and 0.8%), mainly due to gastrointestinal disorders. Even if the transition from MDI to once-daily sc semaglutide in combination with basal insulin were successful in only a minority of patients, the clinical advantage and reduction in burden of disease management that would be associated with transitioning from 3-4 injections of insulin per day to a regimen of once- weekly sc semaglutide and a once-daily injection of basal insulin would be a rather dramatic and remarkable transformation for patients, and one that would likely improve patients' diabetes treatment satisfaction. It would also help to solidify the effectiveness and safety of semaglutide in yet another population of patients with T2D. What cannot be minimized is the tremendous impact that a successful transition to once-weekly semaglutide and once-daily basal insulin could have on patients in terms of reducing their insulin requirements, assisting with weight loss (or mitigating further weight gain), and reducing the frequency and burden of hypoglycemia. In my clinical experience, once patients are titrated to full dose GLP-1RA therapy and attain adequate glycemic control, insulin doses (particularly prandial insulin) can often be further reduced or eliminated without negatively impacting glycemic control. Continuing the insulin therapy at higher doses in these patients simply suppresses the glucose-dependent secretion of endogenous insulin being promoted by the GLP-1RA therapy. Often, only an abrupt cessation of prandial insulin, or a step-wise down-titration of insulin therapy in these patients, will reveal that insulin therapy is no longer required at higher doses to maintain glycemic control. When this does successfully occur, the impact on patients is transformational.

The purpose of this study is to investigate the ability of once-weekly sc semaglutide (in combination with once-daily basal insulin) to maintain or improve glycemic control in patients currently receiving MDI, while providing the patients with a significant reduction in the burden of disease management. In addition, this approach may also furnish a positive effect on weight management, a reduction in hypoglycemic episodes, and improvement in diabetes treatment satisfaction, when substituted for basal/bolus therapy in patients with T2D who currently have adequate glycemic control (A1C ≤ 7.5%) with a regimen of MDI (requiring a total of ≤ 80 units of insulin per day). The A1C cut-point of ≤ 7.5% was chosen because many patients on complex treatment regimens (MDI) with reasonable control, i.e., 7-7.5%, would be expected to have a realistic chance of success by switching from MDI to sc semaglutide and basal insulin combination therapy. Also, many patients taking complex insulin regimens (MDI) fall in the close to A1C goal range of 7-7.5%, so using this cut-point, vs. < 7%, would make recruitment easier. Lastly, patients receiving MDI who are older and/or with heart disease also have higher individual A1C goal/targets around 7.5%. This study will also assess the impact that a successful substitution may have on the patients' diabetes treatment satisfaction, an important, yet under-appreciated aspect of diabetes management.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: men and women
2. Ethnicity: all ethnic groups
3. Language: English
4. Age: ≥ 18 to 75 years
5. Type II diabetes

   * Currently treated with MDI (basal/bolus regimen) for at least 6 months
   * MDI must consist of three or more injections of insulin per day, with at least 2 injections being prandial/rapid-acting insulin
   * Prandial insulin restricted to insulin aspart, glulisine, and lispro
   * Basal insulin restricted to long acting once-daily analogues (insulin glargine U- 100, insulin degludec (U-100 or U-200), or insulin glargine U-300)
   * A1C within 30 days of randomization must be ≤ 7.5% on the present therapy
   * Less than or equal to 120 units of total insulin therapy per day
6. Ability to provide informed consent before any trial-related activities. Trial-related activities are any procedure that would not have been performed during normal management of the subject.

Exclusion Criteria:

1. GAD-65 antibody positive
2. Current glucocorticoid therapy greater than 5 mg of daily prednisone (or equivalent dose of other glucocorticoid)
3. Known or suspected allergy to trial medication(s), excipients, or related products, i.e., GLP-1RA therapy or insulin aspart or insulin degludec.
4. The receipt of any investigational drug within 90 days prior to this trial.
5. Previous participation in this trial (Randomized)
6. Mental incapacity or language barrier (non-English speaking)
7. Use of incretin-based therapies <3 months before inclusion in the study

   * DPP-4 inhibitors sitagliptin, saxagliptin, linagliptin, alogliptin
   * GLP-1RA (exenatide, liraglutide, exenatide LAR, dulaglutide, albiglutide, lixisenatide, semaglutide)
   * GLP-1RA/Basal Insulin combination (IGlarLixi, IDegLira)
8. Present use of oral anti-diabetic agents other than metformin and SGLT-2i. The dose of metformin and/or SGLT-2i must be unchanged and stable for the immediate 3 months prior to baseline.
9. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures
10. Personal or family history of medullary thyroid carcinoma
11. Personal or family history of Multiple Endocrine Neoplasia syndrome type 2
12. History of acute or chronic pancreatitis, severe liver disease or LFT's > 2.5X ULN, or severe disease of digestive tract
13. History of bariatric surgery/procedure (gastric banding, gastric sleeve, or Roux-en-Y)
14. Known elevation of serum calcitonin > 50 ng/L

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Pantalone, DO, Principal Investigator — Staff
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodriguez P, Breslaw N, Xiao H, Bena J, Jenkins K, Isaacs D, Zhou K, Griebeler ML, Burguera B, Pantalone KM; TRANSITION-T2D Investigators. De-intensification of basal-bolus therapy by replacing prandial insulin with once-weekly subcutaneous semaglutide in individuals with well-controlled type 2 diabetes: A single-centre, open-label randomised trial (TRANSITION-T2D). Diabetes Obes Metab. 2025 Feb;27(2):642-651. doi: 10.1111/dom.16057. Epub 2024 Nov 12. PMID 39532398

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Individual participants who were randomized to the two arms of the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 18 | 53
  >=65 years | 5 | 2 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70.1 [62.7 to 72] | 64.7 [54.5 to 69.3] | 68.6 [58.7 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 8 | 25
  Male | 23 | 12 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 39 | 19 | 58
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 27 | 10 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60
Baseline weight (Kg) [Median (Inter-Quartile Range); unit: Kg] | 103.1 [89.6 to 120.6] | 111.6 [86.6 to 122.8] | 104.6 [89.1 to 121.8]
Baseline HbA1c [Median (Inter-Quartile Range); unit: % glycated hemoglobin] | 6.8 [6.2 to 7.2] | 6.9 [6.5 to 7.3] | 6.8 [6.4 to 7.2]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in HbA1C ≤ 7.5%
Description: Mean change in HbA1C ≤ 7.5% from baseline to 26 weeks between the two groups
Time Frame: 26 weeks
Measure: Mean (95% Confidence Interval); unit: % glycated hemoglobin
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin
Number analyzed (Participants) | 40 | 20
% glycated hemoglobin | -0.5 [-0.7 to -0.3] | 0 [-0.3 to 0.3]
Statistical Analysis 1: Comparison: Once-weekly sc Semaglutide Combined With Once-daily Insulin vs MDI Requiring Multiple Daily Injections of Insulin; Linear mixed effect model was conducted for each endpoint to assess mean change at each time point, with time, treatment groups, the interaction of treatment groups and time, and baseline variables included and adjusted in each model. Mean change difference between patients with MDI and those with Semaglutide (MDI - Semaglutide); Test type: Other — p value of contrast difference compared from MDI to Semaglutide group at specific time point, testing whether contrast difference is equal to 0, which means there is no difference between two groups. The determination of statistical significance was made using Bonferroni-adjusted p-value, setting the significance threshold at 0.01 after multiplicity correction; p = 0.009, Bonferroni-adjusted p-value — p value is adjusted for the multiple comparison. The significance threshold is set to 0.01

2. Secondary Outcome: Mean Weight Change
Description: Mean weight change from baseline in body weight at 26 weeks
Time Frame: 26 weeks
Measure: Mean (95% Confidence Interval); unit: Kg
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin
Number analyzed (Participants) | 40 | 20
Kg | -8.6 [-9.6 to -7.6] | 1.4 [0 to 2.8]
Statistical Analysis 1: Comparison: Once-weekly sc Semaglutide Combined With Once-daily Insulin vs MDI Requiring Multiple Daily Injections of Insulin; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bonferroni-adjusted p-value — p value is adjusted for the multiple comparison. The significance threshold is set to 0.01

3. Secondary Outcome: Hypoglycemic Episodes
Description: Recorded for the overall study period
Time Frame: 26 weeks
Measure: Number (95% Confidence Interval); unit: frequency of hypoglycemic episodes
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin
Number analyzed (Participants) | 40 | 20
frequency of hypoglycemic episodes | .7 [.3 to 1.5] | 1.4 [.5 to 3.9]

4. Secondary Outcome: Mean Change From Baseline in A1C
Description: Change from baseline in A1C at week 26
Time Frame: 26 weeks
Measure: Mean (95% Confidence Interval); unit: actual mean A1C change
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin
Number analyzed (Participants) | 40 | 20
actual mean A1C change | -.5 [-.7 to -.3] | 0 [-.3 to .3]

5. Secondary Outcome: Diabetes Treatment Satisfaction Comparison Between Groups
Description: Change from baseline in diabetes treatment satisfaction at week 26
Time Frame: 26 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin
Number analyzed (Participants) | 40 | 20
units on a scale | 18 [15 to 18] | 14 [12.3 to 17.5]

6. Secondary Outcome: Total Daily Insulin Dose
Description: Mean total insulin dose change (U/day) from baseline to week 26
Time Frame: 26 weeks
Measure: Mean (95% Confidence Interval); unit: units per day of total insulin
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin
Number analyzed (Participants) | 40 | 20
units per day of total insulin | -37.3 [-41 to -33.6] | 42.5 [35.8 to 49.1]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Once-weekly sc Semaglutide Combined With Once-daily Insulin | MDI Requiring Multiple Daily Injections of Insulin
All-Cause Mortality (participants affected / at risk) | 0/40 | 1/20
Serious Adverse Events (participants affected / at risk) | 9/40 | 5/20
Other Adverse Events (participants affected / at risk) | 7/40 | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once-weekly sc Semaglutide Combined With Once-daily Insulin (N=40) | MDI Requiring Multiple Daily Injections of Insulin (N=20)
Fever (General disorders) | 1 (1) | 0 (0) — Fever post COVID vaccine, hospitalized for 1 day
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — COVID and COVID vaccine related
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient developed AKI, was admitted to hospital for 4 days with renal function improving but still impaired. Study medication was stopped
Syncopal episode (Nervous system disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Chronic Ulcer (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Ulcer on extremity
Death (General disorders) | 0 (0) | 1 (1) — Patient was discovered to have passed away based on discovering obituary, no note in medical record. Unknown reasons
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once-weekly sc Semaglutide Combined With Once-daily Insulin (N=40) | MDI Requiring Multiple Daily Injections of Insulin (N=20)
Pain (General disorders) | 7 (7) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT04538352/Prot_SAP_000.pdf